CLINICAL TRIAL: NCT05875298
Title: Implementation Of Physical Therapy Protocol In Management Of Chronic Maxillary Sinusitis :A Randomized Controlled Trial
Brief Title: Implementation Of Physical Therapy Protocol In Management Of Chronic Maxillary Sinusitis
Acronym: CRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Saeed Halmy, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003842
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Chronic Maxillary Sinusitis
Keywords: physical therapy protocol; chronic maxillary sinusitis

STUDY DESIGN:
Intervention Model Description: physical therapy protocol and medication
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- physical therapy protocol (Experimental): the patients will receive physical therapy protocol three times a week for four weeks
  Interventions: Other: physical therapy protocol
- physical therapy protocol and medical drugs (Experimental): the patients will receive physical therapy protocol three times a week for four weeks and medication twice daily for four weeks
  Interventions: Other: physical therapy protocol and medical drugs; Other: medical drugs
- medical drugs (Active Comparator): the patients will receive medical drugs twice daily for four weeks
  Interventions: Other: medical drugs

INTERVENTIONS:
Other: physical therapy protocol — the patients will receive physical therapy protocol in the form of therapeutic ultrasound (pulsed mode n An intensity of 1.7 W/cm² for maxillary, respectively in A frequency of 1.7 MHz in Duration of treatment of ten minutes for each maxillary sinus and five minutes for each side), Hot pack that will be applied eight minutes at each maxillary area and manual drainage technique for maxillary sinus.
  Arms: physical therapy protocol
Other: physical therapy protocol and medical drugs — the patients will receive physical therapy protocol and medical drugs in the form of therapeutic ultrasound (pulsed mode n An intensity of 1.7 W/cm² for maxillary, respectively in A frequency of 1.7 MHz in Duration of treatment of ten minutes for each maxillary sinus and five minutes for each side), Hot pack that will be applied eight minutes at each maxillary area and manual drainage technique for maxillary sinus. The drugs will be concentrated sea water 3% and Local corticosteroids nasal spray.
  Arms: physical therapy protocol and medical drugs
Other: medical drugs — The drugs will be concentrated sea water 3% and Local corticosteroids nasal spray.
  Arms: medical drugs; physical therapy protocol and medical drugs

SUMMARY:
this study will be conducted to investigate the effect of physical therapy protocol and medication on pain, pressure pain threshold and dysfunction in patients with Chronic Maxillary Sinusitis

DETAILED DESCRIPTION:
Rhino sinusitis is one of the most common health-care problems worldwide and its prevalence and incidence is increasing. Chronic Sinusitis is a big health problem worldwide that affects almost 15% of humans. The most affected sinus is the maxillary sinus as its drainage orifice through the hiatus semilunaris is badly placed near the roof of the sinus. The first line of treatment for sinusitis is mostly medical drugs including antimicrobial drugs, decongestants, nasal sprays, corticosteroids, and antihistamine drugs which can effectively dry the mucus. Physical therapy also offers a variety of treatment approaches for sinusitis. It includes various electrotherapy modalities, manual drainage techniques, suboccipital release for sinus headaches, needling, and rhino flow therapy. In spite of many studies and treatment approaches done on sinusitis, there are limitations faced in evidence of which approval is most effective, The objective of our study is to investigate the effect of physical therapy protocol in people with chronic maxillary sinusitis.sixty six patients with chronic maxillary sinusitis will be allocated randomly to three groups; one group will receive physical therapy protocol, second one will receive medication only and the third one will receive physical therapy protocol and medication for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* patients clinically diagnosed by ENT Physician with chronic maxillary sinusitis With a history of 3 months or longer.
* Age group from 18 to 50 years

Exclusion Criteria:

* Local contraindications for face mobilization or massage. (abrasions, skin conditions, broken bones) Medical contraindications. (bacterial infections, conjunctivitis, styes)
* Duration of onset less than 2 months Headache due to reasons other than chronic sinusitis (TMJD, cervicogenic headache, underlying neurological diseases, anxiety-related, etc)
* Patients with surgery performed in the past 1 year for maxillary sinusitis Cognition level impairment
* Metal implants in the face region

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  by visual analogue scale (VAS) 10 cm line with 2 ends, 0 and 10 ends 0 end means no pain 10 end means the worst pain
pressure pain threshold | up to four weeks
  pressure algometer will be used to measure pressure pain threshold
functional disability | up to four weeks
  Rhinosinusitis Disability Index will be used to assess functional disability in patients with chronic maxillary sinusitis.it consists of 30 items divided between three main domains: physical, functional, and emotional. Responses are provided using a 5-point Likert scale, and scores range from 0 to 150, with higher scores indicating that CRS exerts a greater impact on quality of life